CLINICAL TRIAL: NCT00947167
Title: A Phase II Study of Pertuzumab and Erlotinib for Metastatic or Unresectable Neuroendocrine Tumors
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Extreme toxicity of Pertuzumab and Erlotinib combination
Sponsor: Pamela L. Kunz (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Pamela L. Kunz, Assistant Professor, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NET0008; SU-03272009-2039; 16186 (Other: Stanford IRB); END0008 (Other: Old OnCore Number)
Record Dates: First submitted 2009-07-23; First posted 2009-07-27 (Estimated); Results first posted 2017-03-03 (Actual); Last update posted 2017-03-03 (Actual); Status verified 2017-01

CONDITIONS: Neuroendocrine Tumors; Carcinoid Tumors; Adrenal Gland Tumors; Neuroblastoma; Pancreatic Neuroendocrine Tumors; Multiple Endocrine Neoplasia
MeSH Terms: conditions — Neuroendocrine Tumors; Carcinoid Tumor; Adrenal Gland Neoplasms; Neuroblastoma; Multiple Endocrine Neoplasia | interventions — pertuzumab; (18F)GTP1; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pertuzumab and Erlotinib (Experimental)
  Interventions: Drug: pertuzumab; Drug: erlotinib

INTERVENTIONS:
Drug: pertuzumab — 840 mg, 420 mg, iv
  Other Names: 2C4; Omnitarg; Genentech
Drug: erlotinib — 150 mg, PO
  Other Names: Tarceva; Erlotinib hydrochloride

SUMMARY:
To determine objective response rates (RR) by RECIST guideline version 1.1 for all patients treated with this strategy consisting of initial therapy with pertuzumab as a single agent and then addition of erlotinib for those who have stable disease or progressive disease at three months (Simon design).

ELIGIBILITY:
Inclusion Criteria:

Subjects must be treated at Stanford University Medical Center for the entire length of study participation.

1. Patients must have histologically or cytologically confirmed well-differentiated neuroendocrine tumor. Patients must be deemed unresectable due to involvement of critical vasculature or adjacent organ invasion or have metastatic disease.
2. Patients with prior surgical resection who develop radiological or clinical evidence of metastatic cancer do not require separate histological or cytological confirmation of metastatic disease unless an interval of > 5 years has elapsed between the primary surgery and the development of metastatic disease. Clinicians should consider biopsy of lesions to establish diagnosis of metastatic disease if there is substantial clinical ambiguity regarding the nature or source of apparent metastases.
3. Prior chemotherapy will be permitted.
4. Prior or concurrent somatostatin analogue use will be permitted.
5. Patients must have a primary or metastatic lesion measurable in at least one dimension by Modified RECIST criteria (v1.1) within 4 weeks prior to entry of study.
6. Patients must have ECOG performance status of 0-2.
7. Patients must be >= 18 years of age.
8. Laboratory values <= 2 weeks prior to randomization:

   * Absolute Neutrophil Count (ANC) >= 1.5 x 109/L (>= 1500/mm3)
   * Platelets (PLT) >= 50 x 109/L (>= 100,000/mm3) (or >= 25 x 109/L (>= 100,000/mm3) if thrombocytopenia is secondary to a non-myelosuppressive cause such as splenic sequestration).
   * Hemoglobin (Hgb) >= 9 g/dL
   * Serum creatinine <= 1.5 x ULN
   * Serum bilirubin <= 1.5 x ULN (<= 3.0 x ULN if liver metastases present)
   * Aspartate aminotransferase (AST/SGOT), alanine aminotransferase (ALT/SGPT) <= 3.0 x ULN (<= 5.0 x ULN if liver metastases present). Note: ERCP or percutaneous stenting may be used to normalize the liver function tests.
   * Albumin >= 1.5
9. LVEF by TTE or MUGA >= 50%
10. Life expectancy >= 12 weeks
11. Ability to give written informed consent according to local guidelines

Exclusion Criteria:

1. Disease-Specific Exclusions

   1. Prior full field radiotherapy <= 4 weeks or limited field radiotherapy <= 2 weeks prior to enrollment. Patients must have recovered from all therapy-related toxicities. The site of previous radiotherapy should have evidence of progressive disease if this is the only site of disease.
   2. Prior biologic or immunotherapy <= 2 weeks prior to registration. Patients must have recovered from all therapy-related toxicities
   3. If history of other primary cancer, subject will be eligible only if she or he has:

      * Curatively resected non-melanomatous skin cancer
      * Curatively treated cervical carcinoma in situ
      * Other primary solid tumor curatively treated with no known active disease present and no treatment administered for the last 3 years
   4. Concurrent use of other investigational agents and patients who have received investigational drugs <= 4 weeks prior to enrollment.
2. General Medical Exclusions

   1. Subjects known to have chronic or active hepatitis B or C infection with impaired hepatic function (ineligible if AST and ALT > 3.0 x ULN).
   2. History of any medical or psychiatric condition or laboratory abnormality that in the opinion of the investigator may increase the risks associated with study participation or study drug administration or may interfere with the conduct of the study or interpretation of study results
   3. Male subject who is not willing to use adequate contraception upon enrollment into this study and for 6 months following the last dose of second-line treatment
   4. Female subject (of childbearing potential, post-menopausal for less than 6 months, not surgically sterilized, or not abstinent) who is not willing to use an oral, patch or implanted contraceptive, double-barrier birth control, or an IUD during the course of the study and for 6 months following the last dose of second-line treatment
   5. Female subject who is breast-feeding or who has positive serum pregnancy test 72 hours prior to randomization
   6. Pleural effusion or ascites that causes respiratory compromise (>= CTCAE grade 2 dyspnea)
   7. Any of the following concurrent severe and/or uncontrolled medical conditions within 24 weeks of enrollment which could compromise participation in the study:

      * Unstable angina pectoris
      * Symptomatic congestive heart failure
      * Myocardial infarction <= 6 months prior to registration and/or randomization
      * Serious uncontrolled cardiac arrhythmia
      * Uncontrolled diabetes
      * Active or uncontrolled infection
      * Interstitial pneumonia or extensive and symptomatic interstitial fibrosis of the lung
      * Chronic renal disease
   8. Patients unwilling to or unable to comply with the protocol
   9. Life expectancy of less than 12 weeks
   10. Current, recent (within 4 weeks of the first infusion of this study), or planned participation in an experimental drug study other than a Genentech-sponsored cancer study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2009-03; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Kunz, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Pertuzumab Alone
Arm/Group | Pertuzumab and Erlotinib
Started | 4
Completed | 4
Not Completed | 0
Period: Erlotinib Added to Pertuzumab
Arm/Group | Pertuzumab and Erlotinib
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Pertuzumab and Erlotinib
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 46.5 [34 to 55]
Gender [Count of Participants; unit: Participants]
  Female | 2
  Male | 2

OUTCOME MEASURES:

1. Primary Outcome: Response Rate (RR) for All Patients Treated With This Strategy (Simon Design)
Description: RECIST v1.1 used
Time Frame: CT scans are done every 4 cycles (every 12 wks)
Population: whole cohort
Measure: Count of Participants; unit: Participants
Arm/Group | Pertuzumab and Erlotinib
Number analyzed (Participants) | 4
Participants | 0

2. Secondary Outcome: Toxicities Assessed by CTCAE Grading Criteria and Assigned Attributions Accordingly
Description: by CTCAE
Time Frame: AEs are assessed every cycle (every 3 wks)
Population: whole cohort
Measure: Count of Participants; unit: Participants
Arm/Group | Pertuzumab and Erlotinib
Number analyzed (Participants) | 4
Participants | 4

ADVERSE EVENTS:
Time Frame: 4 years
Description: We followed patients until death
Arm/Group | Pertuzumab and Erlotinib
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 4/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pertuzumab and Erlotinib (N=4)
Hemoglobin (Blood and lymphatic system disorders) | 3 (3)
Leukocytes (Blood and lymphatic system disorders) | 1 (1)
Platelets (Blood and lymphatic system disorders) | 1 (1)
Fatigue (General disorders) | 4 (4)
Sweating (General disorders) | 1 (1)
Hair loss (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 4 (4)
Anorexia (Gastrointestinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 4 (4)
Mucositis (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2 (2)
Taste (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3)
Hemorrhage (Gastrointestinal disorders) | 1 (1)
Albumin low (Metabolism and nutrition disorders) | 1 (1)
Alkaline Phosphatase elevation (Metabolism and nutrition disorders) | 1 (1)
ALT elevation (Metabolism and nutrition disorders) | 3 (3)
AST elevation (Metabolism and nutrition disorders) | 2 (2)
Calcium low (Metabolism and nutrition disorders) | 1 (1)
Potassium low (Metabolism and nutrition disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination due to toxicity, thus small number of patients analyzed and limited statistical power.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No